CLINICAL TRIAL: NCT01510262
Title: Repeat STI Patients: Tailored Socio-Contextual Intervention to Reduce HIV Risk
Brief Title: Repeat Sexually Transmitted Infection (STI) Patients: Tailored Socio-Contextual Intervention to Reduce HIV Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lance Weinhardt, Professor of Community and Behavioral Health Promotion, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3257547; R01MH089129-01A1 (NIH)
Record Dates: First submitted 2012-01-05; First posted 2012-01-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Sexually Transmitted Infection; HIV
Keywords: Repeat STI patients; HIV; Cost effectiveness; Resource scarce; Urban clinics
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Socio-Contextual Intervention (Experimental): 1. Develop strengths based case management intervention using input from interviews with repeat STI patients, consultants, & piloting.
  2. Recruit/enroll in the intervention 500 subjects (50% women; African American focus).
  3. After subjects receive STI diagnosis, treatment,& partner notification services, randomly assign subjects to:
     A. The STI strengths-based prevention case management, or B. Standard care.
  4. Assess participants' risk behavior, determinants of behavior & quality of life. Investigators will assess the incidence of new STI & test the efficacy of the intervention relative to control.
  5. Conduct a qualitative evaluation. Investigators will sample repeaters and non-repeaters from the experimental group.
  6. Conduct cost effectiveness analyses of intervention compared to the standard.
  Interventions: Behavioral: Tailored Socio-Contextual Intervention
- Standard of Care (Active Comparator): Currently, the total time spent in an STI exam w/men is 30 minutes & 60 w/women. More time is devoted to patients with sexual assault hx. Reason for the visit, symptoms, STI hx, contraception, condom use, number/gender of partners & number/type of sexual activities are assessed. The nurse takes a health hx and asks about typical HIV risks behavior. Due to time the risk assessment is 5 minutes. A risk reduction kit including condoms is issued. Information includes symptoms/treatment of STI, location of sexual health clinics, location of free condoms & testing/treatment resources. Referral information is provided when needed & more involved w/sexual assault survivors. Partner notification is conducted w/syphilis and HIV. This didactic process follows the medical model.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Tailored Socio-Contextual Intervention — 1. Develop strengths based case management intervention using input from interviews with repeat STI patients, consultants, & piloting.
  2. Recruit/enroll in the intervention 500 subjects (50% women; African American focus).
  3. After subjects receive STI diagnosis, treatment,& partner notification services, randomly assign subjects to:
     A. The STI strengths-based prevention case management, or B. Standard care.
  4. Assess participants' risk behavior, determinants of behavior & quality of life. Investigators will assess the incidence of new STI & test the efficacy of the intervention relative to control.
  5. Conduct a qualitative evaluation. Investigators will sample repeaters and non-repeaters from the experimental group.
  6. Conduct cost effectiveness analyses of intervention compared to the standard.
  Arms: Tailored Socio-Contextual Intervention
Behavioral: Standard of Care — Currently, the total time spent in an STI exam w/men is 30 minutes & 60 w/women. More time is devoted to patients with sexual assault hx. Reason for the visit, symptoms, STI hx, contraception, condom use, number/gender of partners & number/type of sexual activities are assessed. The nurse takes a health hx and asks about typical HIV risks behavior. Due to time the risk assessment is 5 minutes. A risk reduction kit including condoms is issued. Information includes symptoms/treatment of STI, location of sexual health clinics, location of free condoms & testing/treatment resources. Referral information is provided when needed & more involved w/sexual assault survivors. Partner notification is conducted w/syphilis and HIV. This didactic process follows the medical model.
  Arms: Standard of Care

SUMMARY:
People who present repeatedly at Sexually Transmitted Infection (STI) clinics represent a key population for HIV prevention intervention research. Despite their heightened risk there is an absence of empirical research on strategies to intervene with repeat STI. Some STI-clinic based behavioral HIV prevention studies, focusing on the general STI patient population, have found that risk reduction interventions can reduce the incidence of a subsequent STI. Studies have shown that expedited treatment for STI patients' partners can reduce subsequent STI and enhancing partner notification can reduce risk for repeat infection. Those who go on to experience repeat infections, after they are provided with risk reduction services, are the focus of this project. Repeat STI literature noted, there have been no intervention studies conducted to lower STI/HIV risk specifically among people who are presenting with repeat STI.

The proposed study develops a risk reduction intervention designed for STI repeaters and evaluates the efficacy of this intervention and its cost-effectiveness. The investigators expect that the intervention for STI repeaters will be significantly more effective than standard care with regard to reducing participants' STI/HIV risks. However, even a highly-effective intervention is unlikely to be adopted if the outcomes come at a high cost. Administrators need to know how effective a "new" intervention is, but also if it is more cost-effective than the program it replaces.

Cost-effectiveness information also is critical to justify the "new" intervention to prevention funders (Milwaukee Department of Health), who are concerned not only with costs and effects, but also with the tradeoff between them. The proposed study will provide the comprehensive level of information about intervention effects and cost-effectiveness required by administrators and resource allocation decision makers to determine whether or not to fund or implement the intervention.

Hypothesis 1. The investigators expect a greater reduction in unprotected vaginal and anal intercourse in the prevention case management compared to the standard care condition.

Hypothesis 2. The hypothesis that the case management group will have a lower STI re-infection rate compared to the standard care group will be tested using each participant's repeat STI status over the 12 month FU period.

DETAILED DESCRIPTION:
This study is a five-year project to develop and test an intervention to reduce risk among people at high vulnerability for HIV infection: patients who present repeatedly at sexually transmitted infection clinics. Repeat bacterial sexually transmitted infections (STI) such as chlamydia, gonorrhea, trichomoniasis, and syphilis, and repeat visits to STI clinics for exposure and potential infection, indicate persistent high-risk sexual behavior. Recidivist patients further represent a significant proportion of public STI clinic visits. Repeat STI can increase the likelihood of HIV transmission during exposure and some recidivist patients may serve as "core transmitters," propagating an ongoing epidemic or endemic chain within a community. Repeat STI patients also face serious health risks from STI complications. In sum, STI repeaters present significant public health risks and place a large financial and resource burden on treatment systems.

Patients with repeat STI, by definition, are not adequately served by the prevention services currently provided by STI clinics. Thus, additional clinic-based services to reduce patients' risk of future infections of STI and HIV are warranted. Adequately addressing the needs of repeat STI patients will allow limited resources to be more heavily invested in services for first-time STI patients who are more likely than recidivist patients to be amenable to standard clinic-based risk-reduction interventions.

The HIV prevention field has largely been silent about assisting patients who present repeatedly with STI and STI risk; there are no published studies testing interventions specifically for repeat STI patients. In addition, most risk-reduction intervention research based in STI clinics has focused directly on the presenting problem of sexual risk behavior or addressed a single co-existing factor (substance use, depression). However, research suggests that repeat STI is related to a wide-ranging and complex configuration of contextual factors that varies by patient. Indeed, repeat STI is highest among communities with the highest rates of STI in general, which are characterized by myriad contextual challenges (unemployment, poverty).

Novel intervention approaches are needed to help repeat STI patients reduce their risk for HIV infection and for infecting others. Investigators propose to address these gaps in the HIV and STI prevention literature by focusing on a high-risk group of recidivist patients: economically disadvantaged urban African Americans. The intervention will help patients address broader, "risk-regulating" social and contextual factors identified by each patient (employment, housing, domestic violence, substance abuse). Investigators also will address individual risk behavior and affective and self-regulatory factors (fatalism, problem solving skills), that contribute to continued risk behavior and interfere with maintenance of risk reduction after an STI.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older;
* Presentation for diagnosis of STI;
* Previous bacterial STI diagnosis in the clinic more than 30 days ago and within the past 12 months;
* No HIV-positive test result in the past; and
* Written informed consent for participation.

Exclusion Criteria:

* Not 18 or older;
* Does not present for STI diagnosis;
* No previous bacterial STI diagnosis in the clinic more than 30 days ago and within the past 12 months;
* HIV-positive test result in the past; or
* No written informed consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
STI Outcome Measures | 12 month follow up visit
  Investigators wish to assess if patients contracted repeat STIs during the study.
  1. Investigators will conduct STI clinic chart abstraction at 12-months post-enrollment to record subsequent episodes of STIs. Because the Milwaukee Health Department electronic STDMIS System includes data from CDC reportable tests conducted elsewhere, investigators will record STIs diagnosed at other sites.
  2. Investigators will test for these STIs and HIV at the 12 month follow up visit.
  3. Investigators will ask patients to report other STI diagnosed anywhere during the period.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline, 4, 8, 12 month follow ups
  Investigators will use the SF-36 version 2 (Quality Metric, 2008) to measure participants' quality of life as a secondary outcome. The 36-item scale assesses eight areas of physical and mental health: physical functioning, impact on physical roles, bodily pain, general health, vitality,social functioning, impacts of emotional factors on social roles, and mental health. The scale and its predecessor, the SF-36, have undergone extensive psychometric development.
Social Action Theory-Based Outcome Mediators | Baseline, 4, 8, 12 month follow ups
  Investigators will assess the action states component of SAT, using a sexual risk reduction specific conceptualization, based on the Information-Motivation-Behavioral Skills model of Fisher & Fisher (1992). Investigators will assess social problem solving style to indicate more general self-regulation skills. Investigators will also assess HIV risk prevention knowledge, HIV risk behavior change motivation, HIV risk reduction skill and self-efficacy, problem solving, life optimism, fatalism, self-esteem, and health related locus of control.
Contextual factors - demographic variables | Baseline, 4, 8, 12 month follow ups
  Demographic variables such as income, housing situation, relationship status, education level, and employment status will be used to characterize participants' economic and social circumstances.
STI Risk Behavior Assessment | Baseline, 4, 8, 12 month follow ups
  Sexual risk behavior will be assessed with a Timeline Followback (TLFB) interview. First, the participant is presented with a calendar and asked to identify days that are personally significant. Second, the investigator defines sex in language understandable & consistent with guidelines. Third, the participant is asked to provide initials of all partners during the reporting period. For each, information is requested (sex; primary, casual, anonymous, HIV positive, IDU, or non-monogamous). Fourth, for each occasion of sexual activity, type of sex, condom use, and AODA are assessed.
Contextual factors - general life context | Baseline, 4, 8, 12 month follow ups
  Social Context Inventory. Investigators will use a list of 54 commonly-experienced social and health issues, adapted from Carey et al., (1999), rated on a scale from 0 (not bothered) to 4 (bothered every day) to identify the salient problems faced by each participant at baseline. Because participants will present with a wide range of challenges beyond the STI, and the SBPCM intervention will focus on helping participants address areas that participants select, this measure will assess progress on goals set in intervention sessions.
Contextual factors - social support | Baseline, 4, 8, 12 month follow ups
  The Social Provisions Scale (Cutrona, 1989) will be used to assess level, type, and satisfaction with available social supports. The global score is the average of 6 subscales: guidance, reliable alliance, worth reassurance, attachment, social integration, and opportunity for nurturance.

CONTACTS AND LOCATIONS:
Overall Officials: Lance S Weinhardt, PhD, Principal Investigator — UW Milwaukee Zilber School of Public Health & Medical College of Wisconsin Center for AIDS Intervention Research
Locations (1):
- University of Wisconsin Milwaukee - Zilber School of Public Health, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Carey MP, Carey KB, Maisto SA, Gordon CM, Weinhardt LS. Assessing sexual risk behaviour with the Timeline Followback (TLFB) approach: continued development and psychometric evaluation with psychiatric outpatients. Int J STD AIDS. 2001 Jun;12(6):365-75. doi: 10.1258/0956462011923309. PMID 11368817
- [Background] Ellen JM, Gaydos C, Chung SE, Willard N, Lloyd LV, Rietmeijer CA. Sex partner selection, social networks, and repeat sexually transmitted infections in young men: a preliminary report. Sex Transm Dis. 2006 Jan;33(1):18-21. doi: 10.1097/01.olq.0000187213.07551.a6. PMID 16385217
- [Background] Ewart CK. Social action theory for a public health psychology. Am Psychol. 1991 Sep;46(9):931-46. doi: 10.1037//0003-066x.46.9.931. PMID 1958012
- [Background] Fortenberry JD, Brizendine EJ, Katz BP, Wools KK, Blythe MJ, Orr DP. Subsequent sexually transmitted infections among adolescent women with genital infection due to Chlamydia trachomatis, Neisseria gonorrhoeae, or Trichomonas vaginalis. Sex Transm Dis. 1999 Jan;26(1):26-32. doi: 10.1097/00007435-199901000-00005. PMID 9918320
- [Background] Golden MR, Whittington WL, Handsfield HH, Hughes JP, Stamm WE, Hogben M, Clark A, Malinski C, Helmers JR, Thomas KK, Holmes KK. Effect of expedited treatment of sex partners on recurrent or persistent gonorrhea or chlamydial infection. N Engl J Med. 2005 Feb 17;352(7):676-85. doi: 10.1056/NEJMoa041681. PMID 15716561
- [Background] Gorsky RD. A method to measure the costs of counseling for HIV prevention. Public Health Rep. 1996;111 Suppl 1(Suppl 1):115-22. PMID 8862166
- [Background] Gunn RA, Fitzgerald S, Aral SO. Sexually transmitted disease clinic clients at risk for subsequent gonorrhea and chlamydia infections: possible 'core' transmitters. Sex Transm Dis. 2000 Jul;27(6):343-9. doi: 10.1097/00007435-200007000-00008. PMID 10907910
- [Background] Hall JM, Stevens PE. Rigor in feminist research. ANS Adv Nurs Sci. 1991 Mar;13(3):16-29. doi: 10.1097/00012272-199103000-00005. PMID 1901470
- [Background] Holtgrave DR, Pinkerton SD. Updates of cost of illness and quality of life estimates for use in economic evaluations of HIV prevention programs. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Sep 1;16(1):54-62. doi: 10.1097/00042560-199709010-00009. PMID 9377126
- [Background] Macias C, Farley OW, Jackson R, Kinney R. Case management in the context of capitation financing: an evaluation of the strengths model. Adm Policy Ment Health. 1997 Jul;24(6):535-43. doi: 10.1007/BF02042831. No abstract available. PMID 9385717
- [Background] Mosack KE, Weinhardt LS, Kelly JA, Gore-Felton C, McAuliffe TL, Johnson MO, Remien RH, Rotheram-Borus MJ, Ehrhardt AA, Chesney MA, Morin SF. Influence of coping, social support, and depression on subjective health status among HIV-positive adults with different sexual identities. Behav Med. 2009 Winter;34(4):133-44. doi: 10.3200/BMED.34.4.133-144. PMID 19064372
- [Background] Orr DP, Johnston K, Brizendine E, Katz B, Fortenberry JD. Subsequent sexually transmitted infection in urban adolescents and young adults. Arch Pediatr Adolesc Med. 2001 Aug;155(8):947-53. doi: 10.1001/archpedi.155.8.947. PMID 11483124
- [Background] Pinkerton SD, Holtgrave DR, DiFranceisco W, Semaan S, Coyle SL, Johnson-Masotti AP. Cost-threshold analyses of the National AIDS Demonstration Research HIV prevention interventions. AIDS. 2000 Jun 16;14(9):1257-68. doi: 10.1097/00002030-200006160-00024. PMID 10894291
- [Background] Weinhardt LS, Galvao LW, Stevens PE, Masanjala WH, Bryant C, Ng'ombe T. Broadening research on microfinance and related strategies for HIV prevention: commentary on Dworkin and Blankenship (2009). AIDS Behav. 2009 Jun;13(3):470-3. doi: 10.1007/s10461-009-9561-y. Epub 2009 Apr 11. No abstract available. PMID 19363651
- [Background] Weinhardt LS, Mosack KE, Swain GR. Development of a computer-based risk-reduction counseling intervention: acceptability and preferences among low-income patients at an urban sexually transmitted infection clinic. AIDS Behav. 2007 Jul;11(4):549-56. doi: 10.1007/s10461-006-9163-x. Epub 2006 Sep 22. PMID 17028993
- [Background] Weinhardt LS, Kelly JA, Brondino MJ, Rotheram-Borus MJ, Kirshenbaum SB, Chesney MA, Remien RH, Morin SF, Lightfoot M, Ehrhardt AA, Johnson MO, Catz SL, Pinkerton SD, Benotsch EG, Hong D, Gore-Felton C; National Institute of Mental Health Healthy Living Project Team. HIV transmission risk behavior among men and women living with HIV in 4 cities in the United States. J Acquir Immune Defic Syndr. 2004 Aug 15;36(5):1057-66. doi: 10.1097/00126334-200408150-00009. PMID 15247559
- [Background] Shain RN, Piper JM, Newton ER, Perdue ST, Ramos R, Champion JD, Guerra FA. A randomized, controlled trial of a behavioral intervention to prevent sexually transmitted disease among minority women. N Engl J Med. 1999 Jan 14;340(2):93-100. doi: 10.1056/NEJM199901143400203. PMID 9887160
- [Background] Hosenfeld CB, Workowski KA, Berman S, Zaidi A, Dyson J, Mosure D, Bolan G, Bauer HM. Repeat infection with Chlamydia and gonorrhea among females: a systematic review of the literature. Sex Transm Dis. 2009 Aug;36(8):478-89. doi: 10.1097/OLQ.0b013e3181a2a933. PMID 19617871
- [Background] Warner L, Klausner JD, Rietmeijer CA, Malotte CK, O'Donnell L, Margolis AD, Greenwood GL, Richardson D, Vrungos S, O'Donnell CR, Borkowf CB; Safe in the City Study Group. Effect of a brief video intervention on incident infection among patients attending sexually transmitted disease clinics. PLoS Med. 2008 Jun 24;5(6):e135. doi: 10.1371/journal.pmed.0050135. PMID 18578564
- [Background] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Background] Cutrona CE. Ratings of social support by adolescents and adult informants: degree of correspondence and prediction of depressive symptoms. J Pers Soc Psychol. 1989 Oct;57(4):723-30. doi: 10.1037//0022-3514.57.4.723. PMID 2795439
- See also: Co-PI's Home Institution — http://www.mcw.edu/cair.htm